CLINICAL TRIAL: NCT02779400
Title: Conformity Measurement Assessment of a Diagnostic Medical Device Used for the Measurement of the INR (International Normalized Ratio)
Brief Title: Assessment of a Diagnostic Medical Device for the INR (International Normalized Ratio) Measurement
Acronym: HEMOPTICS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC/14/54
Record Dates: First submitted 2015-08-27; First posted 2016-05-20 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy; Heart Valves; Arrhythmias, Cardiac; Thromboembolism
Keywords: INR; coagulation; vitamin K antagonist
MeSH Terms: conditions — Arrhythmias, Cardiac; Thromboembolism; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of the device perfomance (Experimental)
  Interventions: Device: Self testing INR device

INTERVENTIONS:
Device: Self testing INR device — the procedure involves a series of repeated measurements of INR with the studied device
  Other Names: In vitro diagnostic device measuring INR

SUMMARY:
The purpose of this study is to assess the measurement conformity of an in vitro diagnostic device measuring the INR (International harmonized Ratio).

DETAILED DESCRIPTION:
The investigators will assess the performance of an in vitro diagnostic device for assessing the INR.

The evaluation will consist of make several INR measurements using the device and compare these measures to the reference value.

The INR will be measured using the study device on capillary blood drops taken from the fingertip. In the same way a venous blood sampling will be carried out to measure a reference INR.

A total of 20 healthy subjects and 180 patients treated with vitamin K agonist will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with vitamin K agonist or healthy volunteers
* For healthy volunteers : Body Mass index between 18 ans 29 kg/m²
* No acute disease in the previous month

Exclusion Criteria:

* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of measurement of the INR with the study device | Just after the blood taken at day 1
  The INR value of each measure with the study device will be compared to the reference INR measured by a central laboratory on a concomitant venous blood sample.

SECONDARY OUTCOMES:
Repeatability of measurement of the INR with the study device | Just after the blood taken at day 1
  Comparison of 8 INR measurements performed with the device in a range of 15 minutes.
Reproductibility of measurement of the INR with the study device | Just after the blood taken at day 1
  Comparison of 8 INR measurements performed with the device in a range of 15 minutes. The modified parameters between measurements will be the lot of consumables and the study device

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research center of Grenoble university hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No